CLINICAL TRIAL: NCT05203172
Title: ENCORAFENIB/BINIMETINIB MASTER PROTOCOL: AN OPEN-LABEL CONTINUATION STUDY FOR PARTICIPANTS CONTINUING FROM ENCORAFENIB/BINIMETINIB CLINICAL STUDIES
Brief Title: The FLOTILLA Study: Providing Continued Access to The Study Medicines Encorafenib and Binimetinib for Participants in Prior Clinical Trials
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4221026; FLOTILLA (Other: Alias Study Number); 2023-509408-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — encorafenib; binimetinib; ribociclib; Cetuximab

STUDY DESIGN:
Intervention Model Description: Each participant will continue to receive the same study treatment regimen at the same dose level as that received in the Parent Studies.
  The details of study intervention and duration of treatment are specified in the applicable Encorafenib/Binimetinib Continuation Sub-Study Protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Binimetinib only treatment (Experimental): For those participants receiving binimetinib treatment in parent studies
  Interventions: Drug: Binimetinib only treatment
- Encorafenib only Treatment (Experimental): For those participants receiving encorafenib only treatment in parent studies
  Interventions: Drug: Encorafenib only Treatment
- Encorafenib & Binimetinib Treatment (Experimental): For those participants receiving encorafenib & binimetinib treatment in parent studies.
  Interventions: Drug: Encorafenib & Binimetinib Treatment
- Treatment of Encorafenib & Binimetinib & Ribociclib (Experimental): For those participants receiving treatment of encorafenib & binimetinib & ribociclib in parent studies
  Interventions: Drug: Treatment of Encorafenib & Binimetinib & Ribociclib
- Treatment of Encorafenib & Binimetinib & Cetuximab (Experimental): For those participants receiving treatment of encorafenib & binimetinib & cetuximab in parent studies
  Interventions: Drug: Treatment of Encorafenib & Binimetinib & Cetuximab

INTERVENTIONS:
Drug: Binimetinib only treatment — Binimetinib will be administered at the same dose level (15 mg to 45 mg) as that received in the Parent Studies C4211001 and C4211003 with water irrespective of food, continuously, starting on Day 1.
  Arms: Binimetinib only treatment
Drug: Encorafenib only Treatment — Encorafenib will be self-administered at the same dose level as that received in the C4221010 Parent Study.
  Arms: Encorafenib only Treatment
Drug: Encorafenib & Binimetinib Treatment — Encorafenib will be administered on a 300 mg QD schedule and binimetinib will be administered on a 45 mg BID schedule, both orally as a flat fixed dose. Cetuximab will be administered at either 400 mg/m2 or 500 mg/m2 IV every 2 weeks on Days 1 and 15 of every cycle.
  Arms: Encorafenib & Binimetinib Treatment
Drug: Treatment of Encorafenib & Binimetinib & Ribociclib — Encorafenib capsule and ribociclib capsules or tablets will be co-administered orally QD with binimetinib tablets BID. The study drugs will be administered as a flat-fixed dose, and not by body weight or body surface area.
  Arms: Treatment of Encorafenib & Binimetinib & Ribociclib
Drug: Treatment of Encorafenib & Binimetinib & Cetuximab — Encorafenib will be administered on a 300 mg QD schedule and binimetinib will be administered on a 45 mg BID schedule, both orally as a flat fixed dose. Cetuximab will be administered at either 400 mg/m2 or 500 mg/m2 IV every 2 weeks on Days 1 and 15 of every cycle.
  Arms: Treatment of Encorafenib & Binimetinib & Cetuximab

SUMMARY:
The purpose of this clinical trial (called the FLOTILLA study) is to give continued access to the study medicines, as well as safety follow-up, for participants in prior clinical trials of encorafenib and/or binimetinib.

All participants who took part in earlier encorafenib and/or binimetinib studies may participate the FLOTILLA study if they are still benefiting from the use of the study medicines. This will be determined by the study doctor. People may not participate in the FLOTILLA study if they have not enrolled in a prior study of encorafenib or binimetinib.

Participants that had enrolled but had stopped receiving the study treatment in a prior study cannot enrolled in this study. Participants in the FLOTILLA study will receive encorafenib and/or binimetinib at the same dose and frequency as in their prior study, for up to about 5 years.

DETAILED DESCRIPTION:
This is an open-label, continuation study for participants receiving study intervention(s) in an encorafenib/binimetinib Parent Study. The study is being conducted under a Master Protocol for Encorafenib/Binimetinib Continuation Sub-Studies with an individual encorafenib/binimetinib continuation sub-study protocol for each eligible Parent Study. Approximately 75 participants from potentially qualifying Parent Studies will be included in this Encorafenib/Binimetinib Continuation study.

This continuation study includes multiple sub-study protocols to allow participants from each of the following parent studies: C4211001 - NCT01320085; C4211003 - NCT01849874; C4221003 - NCT03864042; C4221005 - NCT01543698; C4221006 - NCT03911869; C4221009 - NCT02928224; C4221010 - NCT01436656; C4221013 - NCT02159066; ANCHOR-CRC - NCT03693170

ELIGIBILITY:
Inclusion Criteria:

* Any participant who is receiving study intervention and deriving clinical benefit (as determined by the principal investigator) in an encorafenib/binimetinib Parent Study, with no ongoing NCI CTCAE version 4.03 Grade ≥3 or intolerable Grade 2 AEs considered to be related to study treatment.
* Participants must agree to follow the reproductive criteria as outlined in the applicable Encorafenib/Binimetinib Continuation Sub-Study Protocol.

Exclusion Criteria:

* Any medical reason that, in the opinion of the investigator or sponsor, precludes the participant from inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events leading to permanent discontinuation of study intervention | Baseline up to approximately 5 years
Number serious adverse events reported for all participants | Baseline up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (18):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service Emory University Clinic, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - HealthPartners Cancer Research Center, Saint Paul, Minnesota
  - Regions Hospital Pharmacy, Saint Paul, Minnesota
  - HealthPartners Specialty Center, Saint Paul, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - Rockefeller Outpatient Pavilion (53rd Street), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Investigational Chemotherapy Service, Durham, North Carolina
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Brazil (5):
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo, São Paulo, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo, São Paulo
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Vseobecna fakultni nemocnice v Praze, Prague, Praha 2, Czechia
- France (2):
  - Hopital Claude Huriez - CHU de Lille, Lille, NORD
  - Gustave Roussy, Villejuif, Val-de-marne
- Germany (3):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Otto-von-Guericke-Universitat Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Rambam Health Care Campus, Haifa, Northern District, Israel
- Italy (7):
  - Instituto Tumori Giovanni Paolo II, Bari, Apulia
  - Istituto Nazionale Tumori Regina Elena, Rome, ROMA
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo, Torino
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
- Netherlands (4):
  - Radboudumc, Nijmegen, Gelderland
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, North Holland
  - Nederlands Kanker Instituut Antoni van Leeuwenhoek (NKI AVL), Amsterdam, North Holland
  - Isala, locatie Zwolle, Zwolle
- Portugal (2):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Russia (3):
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg, Sankt-Peterburg
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moscow
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg
- Narodny onkologicky ustav, Bratislava, Bratislava Region, Slovakia
- South Korea (3):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (12):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [LA Coruña]
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Clinic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [lérida]
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
- Lancashire Teaching Hospitals NHS Foundation Trust - Royal Preston Hospital, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221026